CLINICAL TRIAL: NCT00733408
Title: Combined Targeted Therapies for Triple Negative Advanced Breast Cancer - A Phase II Trial of Weekly Nab-Paclitaxel and Bevacizumab Followed by Maintenance Targeted Therapy With Bevacizumab and Erlotinib
Brief Title: Nab-Paclitaxel and Bevacizumab Followed By Bevacizumab and Erlotinib in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Specht, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6628; NCI-2010-00041 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6628 (Other: Fred Hutchinson Cancer Research Center/UW Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Estrogen Receptor-negative Breast Cancer; HER2-negative Breast Cancer; Progesterone Receptor-negative Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tx (chemo, MoAb, and enzyme inhibitor) (Experimental): INDUCTION THERAPY: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients achieving complete response, partial response, or stable disease after completion of induction therapy will receive bevacizumab IV over 30-90 minutes once every 14 or 21 days and erlotinib hydrochloride PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel albumin-stabilized nanoparticle formulation; Biological: bevacizumab; Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774

SUMMARY:
This phase II trial studies how well giving paclitaxel albumin-stabilized nanoparticle (Nab-paclitaxel) formulation together with bevacizumab followed by bevacizumab and erlotinib hydrochloride work in treating patients with metastatic breast cancer. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can prevent cancer growth by blocking the ability of cancer cells to grow and spread. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This trial evaluates a maintenance treatment with erlotinib and bevacizumab after Nab-paclitaxel and bevacizumab which may control cancer growth with biologic therapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Progression free survival.

SECONDARY OBJECTIVES:

I. Response rate.

II. Overall survival.

III. Safety and toxicity.

IV. Exploratory biomarkers will be assessed as potential predictors of response to treatment including: expression of epidermal growth factor receptor (EGFR) and secreted protein acidic and rich in cysteine (SPARC) in the primary tumor and changes in levels of circulating tumor cells (CTCs) and circulating endothelial cells (CECs).

OUTLINE:

INDUCTION THERAPY: Patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients achieving complete response, partial response, or stable disease after completion of induction therapy will receive bevacizumab IV over 30-90 minutes once every 14 or 21 days and erlotinib hydrochloride orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up per physician discretion.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed invasive breast cancer that is estrogen receptor (ER) negative (=< 10%), progesterone receptor (PR) negative (=< 10%) and human epidermal growth factor receptor 2 (HER2) normal (=< 10% of cells) by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH)
* Be receiving first-line therapy for metastatic disease
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) criteria; X-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration; X-rays, scans or other tests for assessment of non-measurable disease must have been performed within 42 days prior to registration
* OR non-measurable disease only, with rising serum cancer antigen (CA)15-3 or CA 27.29 or carcinoembryonic antigen (CEA) documented by two consecutive measurements taken at least 14 days apart with the most recent measurement being within 42 days prior to registration; the second CA 15-3 or CA 27.29 or CEA value must have at least a 20% increase over the first and for CA 15-3 or CA 27.29 be greater than or equal to 40 units/mL or for CEA be greater than or equal to 4 ng/mL
* Subjects with brain metastases as their first site of disease recurrence may be eligible if treated by definitive radiation (stereotactic radiosurgery or whole brain) with clinically controlled neurologic symptoms for a period of 21 days prior to study treatment
* Bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 X upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
* Alkaline phosphatase =< 2.5 X upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
* Platelets > 100,000 cells/mm^3
* Hemoglobin > 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Creatinine =< 1.5 mg/dL is recommended; however, institutional norms are acceptable
* If of childbearing potential must have a negative pregnancy test and use an effective method to avoid pregnancy for the duration of the trial and for at least 6 months after completion of study therapy
* Pre-existing peripheral neuropathy, if present, must be < grade 2 (per Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Patients must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional standards and federal guidelines

Exclusion Criteria:

* Recurrent disease within 12 months after completion of adjuvant chemotherapy containing a weekly taxane
* Central nervous system (CNS) metastases that are symptomatic and/or requiring steroids
* Pre-existing nephritic syndrome
* Serious intercurrent medical or psychiatric illness including serious active infection
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either:

  * Urine protein:creatinine (UPC) ratio >= 1.0 at screening OR
  * Urine dipstick for proteinuria > 2+ (patients discovered to have > 2+ proteinuria on dipstick urinalysis at baseline must have a UPC ratio done that is < 1.0 to be eligible; if the UPC ratio is >= 1.0 then the patient should undergo a 24-hour urine collection which must demonstrate =< 1 g of protein in 24 hours for the patient to be eligible)
* Known hypersensitivity to any component of bevacizumab or to nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-04-23 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Specht, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (17):
- United States (17):
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Yuma Cancer Center, Yuma, Arizona
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Bend Memorial Clinic, Bend, Oregon
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Group Health Cooperative, Redmond, Redmond, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Multicare Medical Oncology Hematology, Tacoma, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Tx (Chemo, MoAb, and Enzyme Inhibitor): INDUCTION THERAPY: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients achieving complete response, partial response, or stable disease after completion of induction therapy will receive bevacizumab IV over 30-90 minutes once every 14 or 21 days and erlotinib hydrochloride PO QD in the absence of disease progression or unacceptable toxicity.
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  bevacizumab: Given IV
  erlotinib hydrochloride: Given PO
Period: Overall Study
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Started | 59
Completed | 55
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 47
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Kaplan-Meier survival curves will be used. A 95% confidence interval for the median PFS will be calculated. A lower bound greater than 8 months would be strong evidence that Nab-Paclitaxel- bevacizumab induction therapy followed by bevacizumab-erlotinib hydrochloride maintenance therapy is superior to paclitaxel and bevacizumab. However, a median PFS of 13 months or greater (regardless of whether the 95% confidence interval for the median extends below 8 months) could also indicate promising results.
Time Frame: Time from date of registration to date of first documentation of progression or symptomatic deterioration or death due to any cause, assessed up to 8 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Number analyzed (Participants) | 55
Months | 9.1 [7.2 to 11.1]

2. Secondary Outcome: Overall Survival
Description: Kaplan-Meier survival curves will be used.
Time Frame: Time from date of registration to date of death due to any cause, assessed up to 8 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Number analyzed (Participants) | 55
Months | 18.1 [15.6 to 21.7]

3. Secondary Outcome: Percentage of Participants With Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 8 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Number analyzed (Participants) | 53
percentage of participants
  Partial Response | 74 [62 to 83]
  Stable Disease | 19 [11 to 30]

4. Secondary Outcome: Incidence of Adverse Events as Assessed by National Cancer Institute CTCAE Version 3.0
Description: Adverse events that meet severity grade 2 or greater will be collected and reported. The number and percent of subjects reporting adverse events (all, severe or worse, serious and related) will be summarized for all patients, and stratified by center and other subgroups of interest.
Time Frame: Up to 30 days after treatment discontinuation
Population: Of the 59 patients enrolled, 4 patients failed to complete a single cycle of induction and considered invaluable and therefore were removed from efficacy analysis. Safety analysis included all 59 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Number analyzed (Participants) | 59
Participants
  Grade 3, 4 Toxicities for Induction | 34
  Grade 3, 4 Toxicities for Maintenance | 14

5. Secondary Outcome: EGFR and SPARC Expression in the Primary Tumor
Time Frame: Up to 8 years
Population: Data published that shows that running assay does not provide useful results
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in Levels of Circulating Tumor Cells
Description: Descriptive statistics, such as mean, standard deviation, and range, will be summarized for circulating tumor cells at baseline and last visit.
Time Frame: Baseline to up to 8 years
Measure: Mean (Standard Deviation); unit: log10 of CTC per mL
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Number analyzed (Participants) | 55
log10 of CTC per mL
  log10(CTC) at baseline | 0.857 (0.854)
  log10(CTC) at last visit | 0.531 (0.756)

7. Secondary Outcome: Changes in Levels of Circulating Endothelial Cells
Description: Descriptive statistics, such as mean and standard deviation, will be summarized for circulating endothelial cells at baseline and last visit.
Time Frame: Baseline to up to 8 years
Measure: Mean (Standard Deviation); unit: log10 of CEC per mL
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
Number analyzed (Participants) | 55
log10 of CEC per mL
  log10(CEC) at baseline | 1.458 (0.491)
  log10(CEC) at last visit | 1.332 (0.574)

ADVERSE EVENTS:
Time Frame: Patients were evaluated for adverse events at each study visit for the duration of their participation in the study and for 30 days after the discontinuation.
Arm/Group | Tx (Chemo, MoAb, and Enzyme Inhibitor)
All-Cause Mortality (participants affected / at risk) | 3/55
Serious Adverse Events (participants affected / at risk) | 5/55
Other Adverse Events (participants affected / at risk) | 52/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tx (Chemo, MoAb, and Enzyme Inhibitor) (N=55)
Infection (Infections and infestations) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tx (Chemo, MoAb, and Enzyme Inhibitor) (N=55)
Neutropenia (Blood and lymphatic system disorders) | 16 (19)
Fatigue (General disorders) | 14 (15)
Neuropathy (Nervous system disorders) | 8 (8)
Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Lymphopenia (Blood and lymphatic system disorders) | 8 (10)
Rash (Skin and subcutaneous tissue disorders) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Infection (Infections and infestations) | 3 (4)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (3)
LFT Abnormality (Hepatobiliary disorders) | 2 (2)
Dermatology other (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Weight loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT00733408/Prot_SAP_000.pdf